CLINICAL TRIAL: NCT06681025
Title: An Observational, Multi-center, Prospective and Retrospective Clinical Study to Evaluate the Performance of the NeuMoDx™ EBV Quant Assay 2.0 on the NeuMoDx™ Molecular Systems in Immunocompromised Transplant Patients
Brief Title: Clinical Performance Evaluation of the NeuMoDx™ EBV Quant Assay 2.0 in Immunocompromised Transplant Patients
Status: Completed | Type: Observational
Sponsor: QIAGEN Gaithersburg, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: SMF-21-2132-1-001
Record Dates: First submitted 2024-10-31; First posted 2024-11-08 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2023-10

CONDITIONS: EBV Viremia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: NeuMoDx EBV Quant 2.0 Assay — The NeuMoDx™ EBV Quant Assay 2.0 is an automated in vitro nucleic acid amplification test for the quantification of Epstein-Barr virus (EBV) DNA in EDTA plasma from immunocompromised transplant patients. Transplant patients are screened for EBV viral load as part of their standard of care. The remaining samples from these in vitro diagnostic nucleic acid amplification tests (NAAT) will be analyzed using the NeuMoDx EBV Quant Assay 2.0 to quantify EBV DNA in EDTA plasma. That result will be compared to a comparator in vitro diagnostic assay to evaluate the performance of the NeuMoDx EBV Quant 2.0 assay.

SUMMARY:
The NeuMoDx EBV Quant Assay 2.0 study is a multi-center, observational clinical investigation designed to evaluate the performance of the NeuMoDx EBV Quant Assay 2.0 in quantifying Epstein-Barr virus (EBV) DNA levels in plasma samples from immunocompromised transplant patients. The study compares the NeuMoDx EBV assay's performance against an FDA-cleared comparator assay under routine clinical use conditions, utilizing both the NeuMoDx™ 96 and NeuMoDx™ 288 Molecular Systems. The aim is to demonstrate the quantitative concordance and clinical utility of the assay in monitoring EBV DNA levels as part of patient management.

DETAILED DESCRIPTION:
This study is an observational, multi-center, open-labeled, prospective, and retrospective clinical evaluation aimed at assessing the performance of the NeuMoDx EBV Quant Assay 2.0 on the NeuMoDx™ 96 and NeuMoDx™ 288 Molecular Systems. Plasma samples are collected from immunocompromised patients undergoing solid organ transplant (SOT) or hematopoietic stem cell transplant (HSCT) who are at risk of EBV infection or reactivation. The study includes both fresh and frozen plasma specimens obtained as part of routine clinical care.

The primary objective is to demonstrate the quantitative concordance of the NeuMoDx EBV assay when compared to the cobas® EBV assay (Roche Diagnostics Corporation) using a predefined set of performance criteria. The study also assesses the equivalence of performance between the two NeuMoDx systems (NeuMoDx™ 96 and NeuMoDx™ 288) in quantifying EBV DNA levels across a range of clinical specimens. Secondary objectives include evaluating the assay's performance across different viral load concentrations and subgroups.

ELIGIBILITY:
Inclusion Criteria:

* Immunocompromised transplant patients (Solid Organ Transplant (SOT) or Hematopoietic Stem Cell Transplant (HSCT)).
* Fresh and frozen plasma specimens derived from whole blood collected with EDTA as an anticoagulant.
* Residual fresh or frozen EDTA plasma specimens obtained from routine testing, including specimens collected from the same subject at different timepoints.
* Sufficient sample volume 1.6- 2.0 ml for testing with 2 assays plus discordant testing.
* EDTA plasma samples have been stored under the following conditions:
* 2-8° C up to 7 days and/or -20° C +/- 2° C or colder for up to 6 months following the separation of plasma from whole blood. Or fresh EDTA plasma samples that have not been stored loaded onto the NeuMoDx™ system immediately after they have been separated from whole blood.
* Frozen samples have not gone through more than two freeze/thaw cycles.

Exclusion Criteria:

* Specimens not collected according to the manufacturer's instructions or study protocol.
* Lack of clear subject identification or label on a residual plasma sample
* Unable to obtain required medical chart information.
* Obvious physical damage to the residual sample.
* Specimens that have remained onboard the NeuMoDx System for longer than 8 hours prior to processing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Standard of care for transplant patients undergoing immuno suppression
Sampling Method: Non-Probability Sample
Enrollment: 1070 (Actual)
Dates: Start 2022-08-31 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
Demonstration that the NeuMoDx™ EBV Quant Assay 2.0 achieves its intended performance during normal conditions of use by the intended user in the intended environment | the primary outcome was assessed a single time after collecting and testing specimens over a 19 month duration
  The concordance of the NeuMoDx™ EBV Quant Assay 2.0 to a comparator's test shall meet these performance metrics with EBV-positive samples within the linear range of the NeuMoDx™ EBV Quant Assay 2.0:
  * Slope (m): 0.9 ≤ m ≤1.1
  * R2 ≥ 0.90, or p-value ≥ 0.05
  Due to the variance in EBV qPCR assays, the Intercept (b) of the linearity fit will be characterized with an anticipated range of -1.0 to +1.0 Log10(IU/mL).
  Percent agreement above the threshold (>LoD/LLoQ) of the reference method shall be > 95%, with the lower confidence interval to be > 80%.
  Percent agreement below the threshold (<LoD/LLoQ) of the reference method shall be > 95%, with the lower confidence interval to be > 90%."

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Johnson, Study Director — QIAGEN Gaithersburg, Inc
Locations (1):
- QIAGEN Gaithersburg, Inc., Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Doseeva V, Mostafa HH, Rhoads D, Relich RF, Garner O, Findeisen P, Eigner U, English A, Johnson S. Performance evaluation of the NeuMoDx EBV Quant Assay 2.0 in Comparison with cobas(R) EBV for epstein-barr virus DNA quantification in immunocompromised patients, a multicenter study. Diagn Microbiol Infect Dis. 2025 Nov;113(3):116956. doi: 10.1016/j.diagmicrobio.2025.116956. Epub 2025 Jun 19. PMID 40578123